CLINICAL TRIAL: NCT05474703
Title: Evaluating the Effects of Levonorgestrel-releasing Intrauterine Device and Dydrogestreone on Quality of Life and Sexual Life in Patients With Abnormal Uterine Bleeding.
Brief Title: Evaluation of the Effects of Levonorgestrel-releasing Intrauterine Device and Dydrogestreone on Quality of Life and Sexual Life in Patients With Abnormal Uterine Bleeding.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principial investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Duphastonversusmirena
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Abnormal Uterine Bleeding
Keywords: Dydrogesterone; Levonorgestrel; Abnormal Uterine Bleeding; Quality of life
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AUK with Dydrogestrone: Patients who applied for abnormal uterine bleeding and received oral dydrogesterone therapy for at least 6 months
  Interventions: Other: SF-36 Scores
- AUK with Levonorgestrel releasing intrauterin device: Patients who applied for abnormal uterine bleeding and were administered levonorgestrel-releasing intrauterine device at least 6 months ago
  Interventions: Other: SF-36 Scores

INTERVENTIONS:
Other: SF-36 Scores — From the electronic database system of our hospital, patients who applied to the gynecology polyclinics of our hospital due to abnormal uterine bleeding between August 2020 and December 2021 and were administered oral dydrogesterone therapy or an intrauterine device releasing levonorgestrel for at least six months were reached using the phone numbers registered in the system.
  The patients were informed about the study conducted by teleconference method, and the patients whose verbal consent was obtained were included in the study. After questioning the patients' sociodemographic characteristics such as age, marital status, educational status, income level, employment status, and obstetric history, the patients received the Short form 36 (P-36), consisting of 36 items; The Quality of Life Scale and the Female Sexual Function Scale (FSFI) composed of 19 items were applied.
  Other Names: FSFI scores

SUMMARY:
This study was retrospectively collected from patients who were diagnosed with abnormal uterine bleeding and received oral dydrogesterone therapy for at least six months or who were administered an intrauterine device containing levonorgestrel at least six months ago, and prospectively Short form 36 (P-36); It covers the comparison of the Quality of Life Scale and the Female Sexual Function Scale (FSFI) by asking over the phone.

DETAILED DESCRIPTION:
This study aimed to apply to the Gynecology and Obstetrics Clinic of Istanbul Health Sciences University Kanuni Sultan Süleyman Training and Research Hospital between August 2020 and December 2021, diagnosed with abnormal uterine bleeding between the ages of 18-45 and receive oral dydrogesterone treatment for at least six months or an intrauterine device releasing levonorgestrel. A total of 171 sexually active female patients who were treated were included. Of the patients participating in the study, 86 comprised two groups of patients who received LNG-IUD, and 85 received oral dydrogesterone treatment.

This study was retrospectively collected from patients who were diagnosed with abnormal uterine bleeding and received oral dydrogesterone therapy for at least six months or who had an intrauterine device containing levonorgestrel at least six months ago, and prospectively Short form 36 (P-36); It covers the comparison of the Quality of Life Scale and the Female Sexual Function Scale (FSFI) by asking over the phone.

Patients outside the age range of 18-45, sexually inactive patients, patients in pregnancy or postpartum, patients with known malignancy history or suspected malignancy, patients with abnormal smear results, patients with bleeding diathesis, patients using drugs that may cause vaginal bleeding, gynecological patients. Patients with any organic pathology that could explain bleeding on examination, patients with levonorgestrel-releasing intrauterine mediator dislocated, and patients who had previously received different treatments for abnormal uterine bleeding were not included.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active patients with abnormal uterine bleeding
* Patients with no known malignancy history or suspected malignancy, patients with average smear results,
* Patients without bleeding diathesis,
* Patients using drugs that may cause vaginal bleeding,

Exclusion Criteria:

* Sexually inactive patients
* Patients in pregnancy or postpartum period,
* Patients with a known history of malignancy or suspected malignancy, patients with abnormal smear results,
* Patients with bleeding diathesis,
* Patients using drugs that may cause vaginal bleeding, patients with any organic pathology to explain the bleeding in gynecological examination
* Patients with a dislocated levonorgestrel-releasing intrauterine device
* Patients who have previously received different treatments for abnormal uterine bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients outside the age range of 18-45, sexually inactive patients, patients in pregnancy or postpartum, patients with known malignancy history or suspected malignancy, patients with abnormal smear results, patients with bleeding diathesis, patients using drugs that may cause vaginal bleeding, gynecological patients. Patients with any organic pathology that could explain bleeding on examination, patients with levonorgestrel-releasing intrauterine mediator dislocated, and patients who had previously received different treatments for abnormal uterine bleeding were not included.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Short Form- 36 scores (SF-36) | 6 months
  The difference in quality of life between the two groups will be evaluated with the SF-36 scale.

SECONDARY OUTCOMES:
The Female Sexual Function Index FSFI scores | 6 months
  Sexual life quality difference between the two groups will be evaluated with the FSFI scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided